CLINICAL TRIAL: NCT00126724
Title: A Phase I/II Study of Repeat Intra-articular Administration of tgAAC94, a Recombinant Adeno-Associated Vector Containing the TNFR:Fc Fusion Gene, in Inflammatory Arthritis Subjects With and Without Concurrent TNF-alpha Antagonists
Brief Title: Study of Intra-articular Delivery of tgAAC94 in Inflammatory Arthritis Subjects
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Targeted Genetics Corporation (Industry)
Responsible Party: Rae Saltzstein, Targeted Genetics Corporation
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13G01; NIH Protocol Number: 0504-705
Record Dates: First submitted 2005-08-02; First posted 2005-08-04 (Estimated); Last update posted 2009-07-29 (Estimated); Status verified 2009-07

CONDITIONS: Arthritis, Rheumatoid; Arthritis, Psoriatic; Ankylosing Spondylitis
Keywords: tgAAC94; Rheumatoid arthritis; Inflammatory arthritis; Arthritis; Gene therapy; AAV
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis, Psoriatic; Spondylitis, Ankylosing; Arthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Active Comparator): 1x10^11 DRP/mL tgAAC94
  Interventions: Genetic: tgAAC94 gene therapy vector
- 2 (Active Comparator): 1x10^12 DRP/mL tgAAC94
  Interventions: Genetic: tgAAC94 gene therapy vector
- 3 (Active Comparator): 1x10^13 DRP/mL tgAAC94
  Interventions: Genetic: tgAAC94 gene therapy vector
- 4 (Placebo Comparator)
  Interventions: Genetic: tgAAC94 placebo

INTERVENTIONS:
Genetic: tgAAC94 gene therapy vector — Single Dose 1x10^11 DRP/mL
  Arms: 1
Genetic: tgAAC94 gene therapy vector — Second dose of 1x10^11 DRP/mL tgAAC94 administered once target joint reaches predetermined criteria for re-injection (on or after Week 12) at the same concentration as initial dose.
  Arms: 1
Genetic: tgAAC94 placebo — placebo
  Arms: 4
Genetic: tgAAC94 gene therapy vector — Single Dose 1x10^12 DRP/mL tgAAC94
  Arms: 2
Genetic: tgAAC94 gene therapy vector — Second dose of 1x10^12 DRP/mL tgAAC94 administered once target joint reaches predetermined criteria for re-injection (on or after Week 12) at the same concentration as initial dose.
  Arms: 2
Genetic: tgAAC94 gene therapy vector — Single Dose 1x10^13 DRP/mL tgAAC94
  Arms: 3
Genetic: tgAAC94 gene therapy vector — Second dose of 1x10^13 DRP/mL tgAAC94 administered once target joint reaches predetermined criteria for re-injection (on or after Week 12) at the same concentration as initial dose.
  Arms: 3

SUMMARY:
The 13G01 clinical trial is a Phase I/II dose escalation study designed to be conducted in adults with inflammatory arthritis who have persistent moderate or severe swelling in one or more joints, without a disease severe enough to warrant a change in regimen for the next three months.

The study will permit subjects who are concurrently on anti-tumor necrosis factor (TNF)-alpha antagonists. For subjects on disease modifying antirheumatic drugs (DMARDs), a stable regimen for inflammatory arthritis for the previous three months, with no changes in doses in the four weeks prior to screening will be required.

The primary objectives are:

1. to evaluate the safety of intra-articular administration of tgAAC94 in subjects currently taking TNF-alpha antagonists, and
2. to evaluate the safety of repeat intra-articular administration of tgAAC94 (gene therapy vector).

DETAILED DESCRIPTION:
tgAAC94 is a recombinant adeno-associated virus serotype 2 (AAV2) vector genetically engineered to contain the cDNA for a human tumor necrosis factor receptor (TNFR)-immunoglobulin (IgG1) Fc fusion (TNFR:Fc) gene. The DNA sequence of TNFR:Fc in tgAAC94 codes for a protein sequence identical to etanercept (Enbrel®). TNF-alpha has been strongly implicated as a major participant in the inflammatory cascade that leads to joint damage and destruction in diseases such as rheumatoid arthritis (RA), psoriatic arthritis (PsA) and ankylosing spondylitis (AS).

Intra-articular delivery of the TNFR:Fc gene (tgAAC94) should result in expression of the secreted protein in the joint space and provide local high concentrations of soluble TNFR:Fc for an extended period of time without requiring frequent administration. Thus, this proposed therapy would be useful in those inflammatory arthritis patients who have a persistently problematic joint despite the use of systemic TNF-alpha blockade or who have a limited number of arthritic joints.

Extensive preclinical studies using rAAV2 containing several different transgenes in a variety of animal models have shown efficient and persistent gene transfer and expression with minimal toxicity. The parent virus (wild-type AAV2) is a naturally occurring, non-replicating virus that depends on a helper virus, such as adenovirus, for replication. The recombinant AAV2 vector is unable to replicate in target host cells because it lacks the AAV genes, whose protein products are also required in trans, for replication and packaging of progeny virus. Extensive epidemiological studies have found AAV2 to be non-pathogenic.

Although there is no cure for arthritis, treatment has been revolutionized by the advent of anti-TNF-alpha therapies. These include etanercept (Enbrel®), infliximab (Remicade®) and adalimumab (Humira®), which consist of soluble TNF receptors, chimeric human-mouse anti-TNF-alpha monoclonal antibodies and fully human anti-TNF-alpha monoclonal antibodies, respectively. Clinical studies have shown these products to improve the signs and symptoms, inhibit the structural damage, and impact functional outcomes in patients with these inflammatory arthritides.

ELIGIBILITY:
Inclusion Criteria:

* Rheumatoid arthritis (RA), psoriatic arthritis (PsA), or ankylosing spondylitis (AS) diagnosed according to established criteria.
* Persistent moderate (grade 2) or severe (grade 3) swelling due to inflammatory arthritis in at least one peripheral joint eligible for injection.
* For subjects with RA, an adequate trial of at least one disease-modifying drug (DMARD) prior to screening.
* For subjects currently on DMARD(s), a stable regimen of inflammatory arthritis for the previous three months, with no changes in doses four weeks prior to screening.
* Age greater than 18 years and less than 75 years at the time of screening.
* Willingness to practice effective birth control measures during the study (through week 36), if male or female of reproductive ability.
* Able to give written informed consent.

Exclusion Criteria:

* Disease severe enough to warrant a change in regimen for inflammatory arthritis in the next three months.
* Discontinuation of etanercept in the past because of safety concerns.
* Current use of anakinra (Kineret®)or abatacept (Orencia®).
* Corticosteroid therapy at doses higher than the equivalent of 10 mg prednisone per day.
* Steroid or hyaluronate injection in the target joint or receipt of an investigational agent less than four weeks prior to screening.
* Class IV ACR functional status (Hochberg et al., 1992).
* Any of the following laboratory values: Hemoglobin <8.5 gm/dL, white blood cell count <3500 per mm cube, platelet <100 K/uL, creatinine >2 mg/dL, bilirubin >2 mg/dL, AST or ALT >2 times the upper limit of normal, or abnormal coagulation profiles (>2 seconds beyond upper range of normal PT or PTT).
* Known HIV infection, known hepatitis C infection, or known positive serologic test for hepatitis B surface antigen.
* Positive PPD, unless previously treated with appropriate prophylaxis.
* Pregnancy or lactation, either at the time of screening or planned in the next 18 months.
* Inflammatory bowel disease, such as Crohn's disease or ulcerative colitis.
* Serious medical disease, such as severe liver or kidney disease, uncompensated congestive heart failure, myocardial infarction within six months, unstable angina, uncontrolled hypertension, severe pulmonary disease or uncontrolled asthma, demyelinating neurological disease, history of cancer (other than cutaneous basal and squamous cell carcinoma) with less than five years documentation of a disease-free state, insulin-dependent diabetes, recurrent opportunistic infections or other concurrent medical condition that, in the opinion of the investigator, would make the subject unsuitable for the study.
* Unlikely to comply with protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2005-08; Primary Completion 2008-10 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Serious adverse events | From time of study drug administration through final study visit
Severe or very severe adverse events | From time of study drug administration through final study visit
Study-drug related adverse events | From time of study drug administration through final study visit

SECONDARY OUTCOMES:
Change in tenderness and swelling of target joint | All scheduled study visits
Time to qualifying for second injection of study drug | Week A12 or 18 or 24
Reduction in disease activity, as measured by American College of Rheumatology (ACR) criteria, Disease Activity Score (DAS) or Assessments in Ankylosing Spondylitis (ASAS) criteria, as applicable | Day A0, Weeks A4, 8, 12, 18, 24, Day B0, Weeks B4, B8, B12, B18, B24, B30, withdrawal
Human tumor necrosis factor receptor (TNFR)-immunoglobulin (IgG1) Fc fusion (TNFR:Fc) protein levels in synovial fluid and serum | Serum: Days A0,7,Weeks A4,12,24, Days B0,7,Weeks 8,12,18,24,30, withdrawal. Synovium: Days A0,4,Weeks A12,24, Day B0,Weeks 4,12,24, withdrawal
Serum anti-adeno-associated virus serotype 2 (AAV2) capsid neutralizing antibodies | Day A0, Weeks A4, 12, 24, Day B0, Weeks B4, 12,24, 30, withdrawal
Joint inflammation and damage on MRI scan | Day A0, Weeks A4, 12, 24

CONTACTS AND LOCATIONS:
Overall Officials: Alison Heald, MD, Study Director — Targeted Genetics Corporation
Locations (22):
- United States (22):
  - Sun Valley Arthritis Center, Glendale, Arizona
  - Catalina Pointe Clinical Research, Inc, Tuscon, Arizona
  - Desert Medical Advances, Palm Desert, California
  - Boling Clinical Trials, Upland, California
  - Denver Arthritis Research Center, Denver, Colorado
  - RASF-Clinical Research Center, Boca Raton, Florida
  - Ocala Rheumatology Research Center, Ocala, Florida
  - Radiant Research Stuart, Stuart, Florida
  - Coeur d'Alene Arthritis Clinic, Coeur d'Alene, Idaho
  - Northwestern Center for Clinical Research, Chicago, Illinois
  - The Arthritis Center, Springfield, Illinois
  - Arthritis and Osteoporosis Center of Maryland, Frederick, Maryland
  - Arthritis Center of Reno, Reno, Nevada
  - United Medical Associates, Johnson City, New York
  - Bone and Joint Hospital Research Dept., Oklahoma City, Oklahoma
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Rheumatic Disease Associates, Willow Grove, Pennsylvania
  - Austin Rheumatology Research, Austin, Texas
  - Arthritis Consultation Center, Dallas, Texas
  - Metroplex Clinical Research Center, Dallas, Texas
  - Radiant Research San Antonio Northeast, San Antonio, Texas
  - Seattle Rheumatology Associates, PLLC, Seattle, Washington

REFERENCES:
- [Derived] Heald AE, Fudman EJ, Anklesaria P, Mease PJ; 13G01 Study Team. Single-joint outcome measures: preliminary validation of patient-reported outcomes and physical examination. J Rheumatol. 2010 May;37(5):1042-8. doi: 10.3899/jrheum.090827. Epub 2010 Mar 15. PMID 20231202
- [Derived] Frank KM, Hogarth DK, Miller JL, Mandal S, Mease PJ, Samulski RJ, Weisgerber GA, Hart J. Investigation of the cause of death in a gene-therapy trial. N Engl J Med. 2009 Jul 9;361(2):161-9. doi: 10.1056/NEJMoa0801066. PMID 19587341
- See also: Sponsor Home Page — http://www.targetedgenetics.com